CLINICAL TRIAL: NCT06756932
Title: A Phase 1 Study to Investigate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BGB-21447 (a Bcl-2 Inhibitor) Combinations for Patients With HR+/HER2- Metastatic Breast Cancer
Brief Title: BGB-21447 (Bcl-2 Inhibitor) Combinations for Adults With Hormone-Receptor Positive (HR+)/Human Epidermal Growth Factor Receptor 2 Negative (HER2-) Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BGB-21447-102; CTR20250114 (Registry Identifier: ChinaDrugTrials)
Record Dates: First submitted 2024-12-24; First posted 2025-01-03 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Hormone-receptor-positive Breast Cancer; HER2-negative Breast Cancer; Metastatic Breast Cancer
Keywords: BGB-21447; BGB-43395; metastatic breast cancer; Bcl-2i; CDK4i
MeSH Terms: conditions — Breast Neoplasms | interventions — Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1A: BGB-21447 + Fulvestrant (Experimental): Sequential cohorts of increasing dose levels of BGB-21447 will be evaluated in combination with fulvestrant.
  Interventions: Drug: BGB-21447; Drug: Fulvestrant
- Part 1B: BGB-21447 + BGB-43395 + Fulvestrant (Experimental): Sequential cohorts of increasing dose levels of BGB-21447 will be evaluated in combination with fulvestrant and BGB-43395.
  Interventions: Drug: BGB-21447; Drug: Fulvestrant; Drug: BGB-43395
- BGB-21447 + Fulvestrant Food Effect Substudy (Experimental): Participants will receive BGB-21447 at the recommended dose with a high-fat meal and under a fasted state in combination with fulvestrant.
  Interventions: Drug: BGB-21447; Drug: Fulvestrant
- Part 2: Dose Expansion, BGB-21447 + Fulvestrant (Experimental): Participants will receive BGB-21447 at the recommended dose(s) for expansion determined in Part 1A in combination with fulvestrant.
  Interventions: Drug: BGB-21447; Drug: Fulvestrant

INTERVENTIONS:
Drug: BGB-21447 — Administered orally.
Drug: Fulvestrant — Administered via intramuscular injection.
Drug: BGB-43395 — Administered orally.
  Arms: Part 1B: BGB-21447 + BGB-43395 + Fulvestrant

SUMMARY:
This is a dose escalation and dose expansion study to assess the safety and tolerability of BGB-21447 (a B-cell leukemia/lymphoma 2 inhibitor, Bcl-2i) in combination with fulvestrant, with or without BGB-43395 (cyclin-dependent kinase 4 inhibitor, CDK4i), in adults with HR+/HER2- metastatic breast cancer.

DETAILED DESCRIPTION:
This new study will check how safe and helpful a potential anticancer drug called BGB-21447 (Bcl-2i) is. This drug will be tested in combination with fulvestrant, with or without BGB-43395 (CDK4i), in adults with metastatic breast cancer.

HR+/HER2- tumors account for approximately 70% of all breast cancers and are responsible for most breast cancer-related deaths. While CDK4/6 inhibitors combined with endocrine therapy have improved outcomes for patients with HR+/HER2- metastatic breast cancer, patients eventually develop progressive disease on these therapies and require new treatments.

BGB-21447 is an oral drug that is highly potent and selectively stops a protein called B-cell lymphoma-2 (Bcl-2). Bcl-2 proteins are often overexpressed in some cancers (like HR+ breast cancer) by keeping the cancer cells from dying. Disrupting this pathway is believed to lead to cell death.

BGB-43395 is an oral drug that selectively stops a protein called cyclin-dependent kinase 4 (CDK4). CDK4 is a type of protein that regulates cell growth and division in your body.

Fulvestrant is a treatment that blocks estrogen receptors and reduces estrogen production. Fulvestrant has been approved to treat hormone receptor positive metastatic breast cancer to help stop the cancer cells from growing.

This combination might be a good way to fight cancer, aiming to give patients the best possible treatment. The study is designed to see if this combination is safe and works well.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed HR+/HER2- metastatic breast cancer. Part 1A and 1B: Participants must have received ≥ 1 prior line(s) of treatment for advanced/metastatic disease, including prior endocrine therapy and CDK4/6 inhibitor in either the adjuvant or advanced/metastatic setting. Part 2: Participants must have received 1-3 prior line(s) of treatment for advanced/metastatic disease, including prior endocrine therapy and CDK4/6 inhibitor in either the adjuvant or advanced/metastatic setting.
* Female participants will be required (either continue ongoing or initiate as soon as feasible) to have ovarian function suppression using gonadotropin-releasing hormone (GnRH) agonists (such as goserelin) or be postmenopausal.
* Male participants may be required to use GnRH agonists when being treated with fulvestrant at the discretion of the investigator.
* Participants must have a stable Eastern Cooperative Oncology Group (ECOG) Performance Status of ≤ 1.
* Adequate organ function.
* Female participants of childbearing potential and nonsterile male participants with female partners of childbearing potential must be willing to use a highly effective method of birth control for the duration of the study and for 7 days after the last dose of BGB-21447, 6 months after the last dose of BGB-43395, and 2 years after the last dose of fulvestrant.
* Food effect substudy only: Participants who are able and willing to fast overnight (≥ 10 hours) and consume a high-fat meal.

Exclusion Criteria:

* Prior Bcl-2 inhibitor exposure. For triplet combination cohorts only: Prior therapy selectively targeting CDK4.
* Known leptomeningeal disease or uncontrolled, untreated brain metastases.
* Any malignancy ≤ 3 years before the first dose of study treatment(s) except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated with curative intent (eg, treated papillary thyroid carcinoma, resected basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix or breast).
* For Part 1B: Uncontrolled diabetes.
* History of hepatitis B or active Hepatitis C infection
* China Only: Untreated chronic hepatitis B or chronic hepatitis B virus (HBV) carriers with HBV DNA > 500 IU/ml (or > 2500 copies/ml) at screening.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 6 months
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), laboratory assessments, and AEs that meet protocol-defined dose-limiting toxicity criteria.
Part 1: Recommended Dose for Expansion (RDFE) of BGB-21447 in combination with fulvestrant and in combination with fulvestrant and BGB-43395 | From first dose of the study drug(s) to 30 days after the last dose or initiation of a new anticancer therapy, whichever occurs first, up to approximately 6 to 9 months
  RDFE of BGB-21447 in combination with fulvestrant and in combination with fulvestrant and BGB-43395 will be determined based upon the maximum tolerated dose (MTD) or maximum administered dose (MAD).
Part 2: Objective Response Rate (ORR) | Approximately 12 months
  ORR is defined as the percentage of participants who had confirmed complete response (CR) or partial response (PR) as assessed by the investigator per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.

SECONDARY OUTCOMES:
Part 1: ORR | Approximately 12 months
  ORR is defined as the percentage of participants who had confirmed CR or PR as assessed by the investigator per RECIST v1.1.
Parts 1 and 2: Duration of Response (DOR) | Approximately 12 months
  DOR is defined as the time from the first determination of an objective response until the first documentation of progression or death, whichever comes first, as assessed by the investigator per RECIST v1.1.
Part 1:Time to Response (TTR) | Approximately 12 months
  TTR is defined as the time from the date of the first dose of study drug to the date of the first CR or PR, as assessed by the investigator per RECIST v1.1.
Part 2: Disease Control Rate (DCR) | Approximately 12 months
  DCR is defined as the percentage of participants with best overall response of a CR, PR, and stable disease.
Part 2: Clinical Benefit Rate (CBR) | Approximately 12 months
  CBR is defined as the percentage of participants who achieve CR, PR, or durable stable disease (stable disease ≥ 24 weeks).
Part 2: Progression-Free Survival (PFS) | Approximately 12 months
  PFS is defined as the time from the date of the first dose of study drug to the date of the first documentation of progressive disease as assessed by the investigator, or death, whichever occurs first. The progressive disease assessment is based on RECIST v1.1.
Part 2: Number of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | From the first dose of study drug(s) to 30 days after the last dose; up to approximately 6 months
  Number of participants with AEs and SAEs, including findings from physical examinations, electrocardiograms (ECGs), and laboratory assessments.
Maximum observed plasma concentration (Cmax) of BGB-21447 and BGB-43395 | Up to approximately 2 months
Time to reach maximum observed plasma concentration (Tmax) of BGB-21447 and BGB-43395 | Up to approximately 2 months
Area under the concentration-time curve (AUC) of BGB-21447 and BGB-43395 | Up to approximately 2 months
Apparent terminal elimination half-life (t1/2) of BGB-21447 and BGB-43395 | Up to approximately 2 months
Food Effect Substudy: AUC of BGB-21447 under fasted and fed state | Up to approximately 2 months
Food Effect Substudy: Cmax of BGB-21447 under fasted and fed state | Up to approximately 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (16):
- United States (4):
  - Hoag Memorial Presbyterian, Newport Beach, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Md Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Australia (6):
  - Saint Vincents Hospital Sydney, Darlinghurst, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Western Health Sunshine Hospital, St Albans, Victoria
  - Linear Clinical Research, Nedlands, Western Australia
- China (6):
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (South), Guangzhou, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - Fudan University Shanghai Cancer Centerpudong, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/